CLINICAL TRIAL: NCT07350863
Title: A Phase I, Single-Arm, Open-Label Clinical Study to Evaluate the Safety and Efficacy of U69 in Patients With Relapsed/Refractory T-Cell Acute Lymphoblastic Leukemia/Lymphoma (T-ALL/LBL)
Brief Title: U69-CART-Cells For R/R T-ALL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Prof., The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SZRTALL02
Record Dates: First submitted 2025-12-23; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory T-lymphoblastic Leukemia/Lymphoma
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low-dose group (Experimental): The investigational product is the CXCR4-enhanced CCR9 Chimeric Antigen Receptor T-Cell Injection (CXCR4/CCR9 CAR-T, U69). The planned doses per cohort are:
  Low Dose Cohort: 1 × 10⁶ CAR-positive T cells per kg of body weight. The product is administered as a single intravenous infusion. The actual administered dose is acceptable within a range of 70% to 130% of the target dose. The required cell number will be calculated based on the subject's body weight at the time of apheresis. The Investigator may adjust the final cell dose based on the subject's specific clinical condition.
  Interventions: Drug: CXCR4 CCR9 CAR-T
- Medium dose group (Experimental): The investigational product is the CXCR4-enhanced CCR9 Chimeric Antigen Receptor T-Cell Injection (CXCR4/CCR9 CAR-T, U69). The planned doses per cohort are:
  Medium Dose Cohort: 3 × 10⁶ CAR-positive T cells per kg of body weight. The product is administered as a single intravenous infusion. The actual administered dose is acceptable within a range of 70% to 130% of the target dose. The required cell number will be calculated based on the subject's body weight at the time of apheresis. The Investigator may adjust the final cell dose based on the subject's specific clinical condition.
  Interventions: Drug: CXCR4 CCR9 CAR-T
- High dose group (Experimental): The investigational product is the CXCR4-enhanced CCR9 Chimeric Antigen Receptor T-Cell Injection (CXCR4/CCR9 CAR-T, U69). The planned doses per cohort are:
  High Dose Cohort: 6 × 10⁶ CAR-positive T cells per kg of body weight. The product is administered as a single intravenous infusion. The actual administered dose is acceptable within a range of 70% to 130% of the target dose. The required cell number will be calculated based on the subject's body weight at the time of apheresis. The Investigator may adjust the final cell dose based on the subject's specific clinical condition.
  Interventions: Drug: CXCR4 CCR9 CAR-T

INTERVENTIONS:
Drug: CXCR4 CCR9 CAR-T — CXCR4-enabled CCR9 chimeric antigen receptor T-cell injection solution

SUMMARY:
Overall Introduction This single-arm, open-label clinical trial aims to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of CXCR4-enabled CCR9 chimeric antigen receptor T-cell injection (CXCR4 CCR9 CAR-T) in patients with relapsed or refractory T-lymphoblastic leukemia/lymphoma (r/r T-ALL/LBL). Additionally, the study seeks to preliminarily assess the efficacy of CXCR4 CCR9 CAR-T cells and explore the appropriate dosage and administration schedule for subsequent Phase II clinical trials. A dose escalation study following the 3+3 design was implemented across three dose cohorts, with each cohort planned to enroll 3 to 6 patients, totaling 9 to 18 participants. Following cell infusion, subjects underwent safety and efficacy follow-up, which continued until 2 years post-infusion, subject withdrawal, or study termination-whichever occurred first. For subjects with available follow-up information after study completion or early termination, long-term follow-up-including long-term safety monitoring-was conducted for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be eligible for the study:

  1. Informed Consent: Voluntary provision of written informed consent and anticipated ability to complete all required study procedures and follow-up assessments.
  2. Age: ≥15 and ≤75 years of age at the time of signing the informed consent form.For minors (age ≤ 18 years), informed consent must be provided by a legal guardian; minors with capacity to sign should co-sign the consent form alongside their guardian.
  3. Diagnosis and Disease Status: Histologically or cytologically confirmed diagnosis of relapsed or refractory T-cell acute lymphoblastic leukemia/lymphoma (T-ALL/LBL) according to the 2022 WHO Classification of Haematolymphoid Tumours, for which standard curative treatments are no longer effective.

     3.1 For T-ALL: Presence of ≥5% blasts in bone marrow or peripheral blood at screening. Relapse: Defined as recurrence of blasts (≥5%) in peripheral blood or bone marrow or emergence of extramedullary disease after prior achievement of complete remission (CR/CRi). This includes early relapse (within 12 months of first remission), late relapse (≥12 months) failing to achieve remission after one multi-agent re-induction chemotherapy cycle, or relapse after autologous or allogeneic hematopoietic stem cell transplantation (HSCT).

     Refractory: Defined as failure to achieve CR after at least two cycles of induction chemotherapy, or failure to achieve CR after one cycle of salvage therapy following relapse.

     3.2 For T-LBL: Presence of at least one measurable lesion at screening, defined as a nodal lesion with a long axis >15 mm or an extranodal lesion with a long axis >10 mm, as assessed by CT or MRI per the 2014 Lugano criteria.

     Relapsed/Refractory: Defined as relapse or disease progression after at least two prior lines of therapy; primary refractory disease (failure to achieve at least a partial response, PR, after first-line therapy); or relapse/progression after autologous or allogeneic HSCT (must be confirmed by tissue biopsy).
  4. Biomarker: Confirmed CCR9 positivity on tumor cells via flow cytometry of bone marrow samples and/or via immunohistochemistry of extramedullary lesion biopsies at screening.
  5. Performance Status: Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
  6. Life Expectancy: Estimated life expectancy of greater than 3 months.
  7. Bone Marrow Reserve: Adequate bone marrow reserve at screening, defined as:

     Absolute Neutrophil Count (ANC) ≥ 1.0 × 10⁹/L Absolute Lymphocyte Count (ALC) ≥ 0.3 × 10⁹/L Platelet Count (PLT) ≥ 20 × 10⁹/L (transfusion support is permitted).
  8. Organ Function: Adequate organ function defined as:

     Hepatic: Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 3 × Upper Limit of Normal (ULN); Total Bilirubin ≤ 2 × ULN.

     Renal: Serum Creatinine ≤ 1.5 × ULN, OR Creatinine Clearance ≥ 50 mL/min (calculated by the Cockcroft-Gault formula).

     Cardiac: Left Ventricular Ejection Fraction (LVEF) ≥ 45%. Pulmonary: Oxygen saturation ≥ 92% on room air.
  9. Contraception: Female subjects of childbearing potential must have a negative serum pregnancy test at screening and agree to use highly effective contraception for at least one year post-infusion. Male subjects with female partners of childbearing potential must agree to use barrier contraception and refrain from sperm donation for at least one year post-infusion.
  10. Leukapheresis: Must have adequate venous access for leukapheresis or venous blood draw and no other contraindications to leukapheresis.

Exclusion Criteria:

* Subjects will be excluded from the study if they meet any of the following criteria:

  1. Diagnosis of any other malignancy within 3 years prior to screening, except for those who have completed curative therapy and achieved over 3 years of disease-free survival with a low risk of recurrence as determined by the investigator (e.g., carcinoma in situ of the lung, basal cell carcinoma of the skin).
  2. History or presence of central nervous system (CNS) disorders unrelated to the disease under study at screening or previously, such as seizure, cerebral ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving the CNS.
  3. Prior receipt of cell therapies targeting CCR9, including but not limited to CAR-T or CAR-γδT cells.
  4. Significant or active parenchymal CNS or cranial nerve lesions where, in the investigator's judgment, the risks outweigh the benefits.
  5. Systemic corticosteroid use discontinued ≤72 hours prior to apheresis, except for physiological replacement doses (e.g., prednisone <10 mg/day or equivalent).
  6. Donor lymphocyte infusion (DLI) within 6 weeks prior to apheresis.
  7. Treatment with any anti-T-cell antibody therapy within 4 weeks prior to apheresis.
  8. Presence of any of the following: positive hepatitis B e antibody (HBe-Ab) and/or hepatitis B core antibody (HBc-Ab) with HBV-DNA above the lower limit of quantification; positive hepatitis C antibody (HCV-Ab) with HCV-RNA above the lower limit of quantification; positive treponema pallidum antibody (TP-Ab); positive human immunodeficiency virus (HIV) antibody test; or EBV-DNA or CMV-DNA levels above the lower limit of quantification by quantitative PCR.
  9. Active or uncontrolled infection requiring systemic therapy at the time of screening (excluding mild genitourinary or upper respiratory tract infections), as assessed by the investigator.
  10. Coronary angioplasty or stent placement within 12 months prior to informed consent; congestive heart failure of New York Heart Association (NYHA) Class III-IV; myocardial infarction, unstable angina, or other clinically significant cardiac conditions within 6 months deemed ineligible by the investigator; QTc interval >480 ms (calculated using Fridericia's formula) at screening; or uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg) or pulmonary hypertension despite standard treatment.
  11. Unstable systemic diseases per investigator judgment, including but not limited to severe hepatic, renal, or metabolic diseases requiring pharmacological intervention.
  12. Active or uncontrolled autoimmune disease, or primary/secondary immunodeficiency.
  13. History of severe immediate hypersensitivity to any drug used in the study.
  14. Administration of any live vaccine within 6 weeks prior to screening.
  15. Pregnant or lactating individuals.
  16. History of autoimmune disease requiring systemic immunosuppressive or disease-modifying medication within the past 2 years (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus).
  17. Allogeneic hematopoietic stem cell transplantation within 12 weeks prior to apheresis; presence of acute or moderate-to-severe chronic GVHD within 4 weeks prior to screening; or any systemic GVHD treatment within 4 weeks prior to cell infusion, including those requiring concomitant corticosteroid use.
  18. Participation in any other interventional clinical trial within 4 weeks prior to screening.
  19. Inability to comply with study procedures, or any other condition considered by the investigator to render the subject unsuitable for the study.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Within 28 days after CXCR4 CCR9 CAR-T cell infusion
  DLT refers to any of the following conditions occurring within 28 days after cell reinfusion that are related to cell infusion:
  ① Hematologic DLT: Grade 4 toxicity (excluding lymphopenia) not caused by the underlying disease and taking more than 30 days to resolve to ≤ Grade 2.
  ② Non-hematologic DLT: Any toxicity ≥ Grade 4 that is possibly related to CAR-T therapy, or Grade 3 toxicity that requires ≥7 days to resolve to ≤ Grade 2 or to return to baseline.
Adverse Event (AE） | 2 years
  Record the types, occurrence frequency and severity of adverse events (AEs) related to CAR-T, with specific definitions determined according to CTCAE v5.0.The CRS and ICANS ratings do not use CTCAE but adopt the evaluation criteria in the ASTCT standards.
The Recommended Phase II Dose（RP2D） | Within 28 days after CXCR4 CCR9 CAR-T cell infusion
  The dose recommended for use in phase 2 studies on the basis of dose limiting toxicities observed in phase 1 studies.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 28 days and within 3 months after infusion of CXCR4 CCR9 CAR-T cells
  Defined as the proportion of subjects achieving an objective response (complete or partial response). All subjects not meeting the objective response criteria as of the data cutoff date will be considered non-responders.
  ①For T-ALL patients: Treatment response is defined as the achievement of either Complete Remission (CR) or Complete Remission with Incomplete Hematologic Recovery (CRi);
  ②For T-LBL patients: Treatment response is defined as the achievement of either Complete Response (CR) or Partial Response (PR);
MRD-negative rate (for T-ALL) | 28 days and within 3 months after infusion of CXCR4 CCR9 CAR-T cells
  The proportion of T-ALL patients with negative MRD in the bone marrow when the therapeutic effect reaches remission. T-ALL patients have residual leukemia cells in the bone marrow detected by flow cytometry below 10-⁴ and/or negative qualitative or quantitative detection of bone marrow fusion genes (if any).
Duration of Response (DOR) | 2 years
  It refers to the period from the time when the subject first achieves remission to the time of disease progression or death due to the disease. Subjects who have not experienced disease progression or death by the time of the final data collection will be censored at the time of their last valid tumor assessment. Common reasons for censoring include, but are not limited to:
  * Loss to follow-up; ②Withdrawal from the study; ③Initiation of a new anticancer therapy.
Progression-Free Survival (PFS) | 2 years
  Defined as the time from the date of cell infusion to the date of first documented disease progression or death from any cause, whichever occurs first. Subjects who have not experienced disease progression or death by the data cutoff date will be censored at the time of their last tumor assessment.
Event-Free Survival (EFS) | 2 years
  Defined as the time from the date of cell infusion to the occurrence of any of the following events (whichever comes first):
  * Death from any cause after achieving remission ②Disease relapse or progression ③Treatment failure, defined as either lack of efficacy or discontinuation of the clinical trial due to:
    * Death
    * Adverse events
    * Lack of efficacy or disease progression
    * Initiation of new antitumor therapy
Overall Survival (OS) | 2 years
  Defined as the time from the date of cell infusion to the date of death from any cause. For subjects who are still alive at the time of analysis, OS will be censored on the date of last known contact. It is specifically noted that subsequent allogeneic hematopoietic stem cell transplantation or receipt of any new antitumor therapy will not constitute a censoring event for OS analysis.
Pharmacokinetics-AUC(0-28) | 2 years
  The area under the curve from 0 to 28 days for the reinfusion.
Pharmacokinetics-Cmax | 2 years
  The peak concentration of the drug in the peripheral blood sample.
Pharmacokinetics-Tmax | 2 years
  The time at which the peak concentration of the drug is reached in the peripheral blood sample.
IL-6 | Within 28 days after CXCR4 CCR9 CAR-T cell infusion
  Changes in the levels of IL-6.
IFNγ | Within 28 days after CXCR4 CCR9 CAR-T cell infusion
  Changes in the levels of IFNγ.
Ferritin | Within 28 days after CXCR4 CCR9 CAR-T cell infusion
  Changes in the levels of Ferritin.
C-reactive protein(CRP) | Within 28 days after CXCR4 CCR9 CAR-T cell infusion
  Changes in the levels of CRP.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Baseline characteristics of patients, outcomes
Supporting Information: SAP, CSR
Time Frame: one year after the study termination
Access Criteria: Clinical researchers worldwide can access the IPD and supporting information after author authorization. They can get IPD details by visiting the ResMan system.
URL: http://www.medresman.org.cn/login.aspx

REFERENCES:
- [Background] Li YR, Zhu Y, Chen Y, Yang L. The clinical landscape of CAR-engineered unconventional T cells. Trends Cancer. 2025 Jun;11(6):520-539. doi: 10.1016/j.trecan.2025.03.001. Epub 2025 Mar 27. PMID 40155286
- [Background] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753